CLINICAL TRIAL: NCT06762262
Title: Effects of Pilate Training Versus Moderate Intensity Continous Training on Dyspnea and Cardiovascular Fitness in Hypertensive Patients
Brief Title: Effects of Pilate Training Versus Moderate Intensity Continous Training in Hypertensive Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rabbia Naseer Ahmed
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Prehypertension
Keywords: Hypertension, Dyspnea, Pilates Training, Modified-Intensity Training
MeSH Terms: conditions — Prehypertension; Hypertension; Dyspnea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Moderate-Intensity continuous training (MICT) refers to a type of aerobic exercise that involves maintaining a steady and moderate level of physical activity for an extended period. The exercise is performed at a consistent and moderate pace without significant fluctuations in intensity. MICT primarily targets the aerobic energy system, enhancing cardiovascular endurance and respiratory efficiency
  Interventions: Combination Product: Moderate-Intensity continuous training
- Controlled (Other): Will receive Pilates exercises, Mild stretching, Glute Bridge, Isometric Glute Bridge, Single Leg Raise, Upper Abdominal Curl, Single- leg Strech, Double-Leg Strech, Plank Push Backs, roll down, Cool down. Pilates exercises emphasize controlled movements, proper breathing, and the engagement of the deep core muscles. Pilates exercises can be performed on a mat or using specialized equipment such as a reformer.
  Interventions: Combination Product: Moderate-Intensity continuous training

INTERVENTIONS:
Combination Product: Moderate-Intensity continuous training — refers to a type of aerobic exercise that involves maintaining a steady and moderate level of physical activity for an extended period. The exercise is performed at a consistent and moderate pace without significant fluctuations in intensity. MICT primarily targets the aerobic energy system, enhancing cardiovascular endurance and respiratory efficiency

SUMMARY:
Hypertension, commonly known as high blood pressure, continues to be the leading cause of both sickness and mortality globally. Generally, individuals in good health might have trouble breathing solely during vigorous exercise or when holding their breath, finding relief by stopping the activity or adjusting their breathing technique. Often patients with hypertension seek various treatments to relieve symptoms. The aim of this study is to compare the effects of Pilates Training and Moderate Intensity Continuous Training on dyspnea and cardiovascular fitness in hypertensive patients. The study would be randomized clinical trial. A total of thirty-four subjects will be assigned randomly by using block randomization into two groups. Group A will be given Pilates training while Group B will moderate intensity training. After confirmation of diagnosis with medical history and physical examination as well as chronic, mild-to moderate, and stable (>1 year duration) hypertension (systolic blood pressure [SBP] between 140-179 mm Hg and diastolic blood pressure [DBP]between 90-109 mm Hg) recommended. 3-minute step test, VO2max and Modified BORG scale would be used as an outcome measure tools for cardiovascular parameters and dyspnea. The collected data will be analyzed in SPSS 25.0. Descriptive and inferential statistics will be applied after testing normality of data

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 45 to 70 years old
* Gender: Male and Female both
* Chronic, mild-to moderate, and stable (>1 year duration) hypertension (systolic blood pressure
* [SBP] between 140-179 mm Hg and diastolic blood pressure [DBP] between 90-109 mm Hg).
* Single antihypertensive medication will be recruited.
* Participants have sedentary life style.
* Smokers, alcoholic, diabetic, and other cardiac problems (controlled) would be included.

Exclusion Criteria:

* Patients with Permanent atrial fibrillation
* Patients with COPD
* Patients with Heart surgery
* Patients with presence of symptomatic congestive heart failure
* Smokers, alcoholic, diabetic, and other cardiac, renal, and respiratory disease patients (uncontrolled) would be excluded.
* Participants with no history of psychiatry or psychological disorders or abnormalities.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
6 MWT | 8 weeks
VO2 max | 8 weeks
Borg Dyspnea Scale | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sumera Nassser, Mphill, Study Chair — Riphah International University
Locations (1):
- Sheikh Zaid Hospital, Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: No